CLINICAL TRIAL: NCT00593164
Title: Clinical Study of the LRS ThermoSuit™ System in Post Arrest Patients With Intravenous Infusion of Magnesium Sulfate
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding for study is currently unavailable.
Sponsor: Life Recovery Systems (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LRS-01-07-02
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Death, Sudden, Cardiac; Coma
Keywords: Hypothermia, Induced; Death, Sudden, Cardiac; Resuscitation; Coma
MeSH Terms: conditions — Death, Sudden, Cardiac; Coma; Hypothermia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Comatose post-resuscitation patients cooled with ThermoSuit and treated with intravenous magnesium sulfate (30 mg per kg IV over 15 min).
  Interventions: Device: Cooling with ThermoSuit with Magnesium Sulfate Infusion
- 2 (Active Comparator): Comatose post-resuscitation patients cooled with ThermoSuit and treated with intravenous normal saline.
  Interventions: Device: Cooling with ThermoSuit with Normal Saline Infusion

INTERVENTIONS:
Device: Cooling with ThermoSuit with Magnesium Sulfate Infusion — Cooling with LRS ThermoSuit within 15 minutes of intravenous Magnesium Sulfate infusion (30 mg/kg, added to 100 ml normal NaCl solution, given over 15 min).
  Arms: 1
Device: Cooling with ThermoSuit with Normal Saline Infusion — Cooling with LRS ThermoSuit within 15 minutes of normal saline infusion (100 ml of normal NaCl solution, given over 15 min).
  Arms: 2

SUMMARY:
This study will involve the use of therapeutic hypothermia. This prospective cohort pilot study will evaluate the clinical performance of a new device, the ThermoSuit™ System, to achieve therapeutic hypothermia in comatose patients following resuscitation from cardiac arrest, and the impact of the vasodilator, magnesium sulfate, on cooling performance and hemodynamics in these patients. The study hypothesis is that magnesium sulfate will significantly increase the rate of cooling.

DETAILED DESCRIPTION:
This study will involve the use of therapeutic hypothermia, an accepted medical treatment recommended for comatose post resuscitation patients by the International Liaison Committee on Resuscitation (ILCOR), the American Heart Association (AHA), and the European Resuscitation Council. This prospective cohort pilot study will evaluate the clinical performance of a new device, the ThermoSuit™ System, to achieve therapeutic hypothermia in comatose patients following resuscitation from cardiac arrest, and the impact of the vasodilator, magnesium sulfate, on cooling performance and hemodynamics in these patients. 14 patients will be prospectively randomized to receive either magnesium sulfate or normal saline (placebo) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest prior to or during hospital admission, with restoration/return of spontaneous circulation (ROSC).
* Estimated or known age > 18 years.
* Intubation, ventilation and placement of esophageal temperature probe.
* Persistent neurologic dysfunction i.e. comatose upon enrollment [GCS ≤ 8].

Exclusion Criteria:

* Height greater than 188 cm.
* Elbow-to-elbow width greater than 60 cm (as measured above the supine patient).
* Core temperature less than 35°C after ROSC (as measured in the esophagus).
* Comatose state before the cardiac arrest due to the administration of drugs that depress the central nervous system.
* Known pregnancy.
* Known terminal illness that preceded the arrest.
* Known enrollment in another study of a device, drug, or biologic.
* Major trauma or other co-morbidity requiring urgent surgery.
* > 4 hours since return of spontaneous circulation.
* Severe coagulopathy (with active bleeding).
* Hemodynamic instability despite vasopressors (SBP < 90 mmHg or MAP < 60 mmHg for > 30 minutes after ROSC and before enrollment).
* Bradycardia (HR<60/min)
* Allergy against MgSO4
* AV-block
* Myasthenia gravis
* Known terminal renal insufficiency (creatinine-clearance < 20ml/min)
* Severe myocardial dysfunction (EF<25%)
* Chronic digitalis therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Cooling rate from start of cooling until a temperature of 34°C is reached | Approximately 10 to 60 minutes after start of cooling

SECONDARY OUTCOMES:
Time from collapse to a core temperature < 34.0°C | Approximately 30 to 180 minutes
Percentage of time of the maintenance phase where the patient core temperature is between 32.0 and 34.0°C. | Approximately 12 hours after initial cooling
Incidence of shivering during cooling and maintenance of hypothermia | Approximately 12 hours after cooling
Duration of maintenance of hypothermia without supplemental cooling | Approximately 12 hours after cooling
Total number of days in ICU | Generally less than 30 days
Neurologic and physical status | At discharge, 30 +/- 7 days, and 6 months +/- 15 days after initial treatment
Adverse events, serious adverse events, device-related adverse events | From enrollment through 6-month follow-up
Blood pressure and ECGs | Through hospital stay
Serum chemistry parameters (standard chemistry panel) | Through hospital stay
Hematology parameters | Through hospital stay
Survival | To 24 hours, hospital discharge, and 30 days
Rate of infection (respiratory, skin, and invasive access sites) and rate of sepsis | During hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Holzer, M.D., Principal Investigator — Department of Emergency Medicine, Medical University of Vienna
Locations (1):
- Department of Emergency Medicine, Medical University of Vienna, Vienna, Austria